CLINICAL TRIAL: NCT06851000
Title: The Effects of Ultrasound-guided Pulsed Radiofrequemcy Versus Dry Needling in Myofascial Pain Patients
Brief Title: The Effects of Ultrasound-guided PRF Versus DN in Myofascial Pain Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, Principal investigator, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRF-DN
Record Dates: First submitted 2025-02-13; First posted 2025-02-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Myofascial Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF-PRF (Experimental)
  Interventions: Procedure: ultrasound-guided pulsed radiofrequency
- DN-PRF (Active Comparator)
  Interventions: Procedure: ultrasound-guided dry needling

INTERVENTIONS:
Procedure: ultrasound-guided pulsed radiofrequency — Medication: 0-3months; Pulsed radiofrequency: week 2, 6, 10;
  Arms: PRF-PRF
Procedure: ultrasound-guided dry needling — Medication: 0-3 months; Dry needling: week 2; Pulsed radiofrequency: week 6, 10;
  Arms: DN-PRF

SUMMARY:
This study aims to compare the effects of pulsed radiofrequency and drying needling and explore the short-term effect of pulsed radiofrequency in treating myofascial pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, gender unlimited.
* Myofascial pain diagnosed according to the "Simons and Travell" criteria.
* Able to complete treatment and follow-up.
* Signed inform consent form.

Exclusion Criteria:

* History of surgery, trauma, or infection in the pain area.
* Severe systemic disease, e.g. malignant tumor; severe hepatic, renal, or coagulation disorder; etc.
* Pregnancy, needle phobia, unable to cooperate.
* Concurrently receiving pain treatment in other institutions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Change of mechanical pain threshold (△MPT) | week 0 to week 4
  Mechanical pain threshold was measured by an ergometer called Microfet3. △MPT=MPT4wk (MPT measured at week 4)-MPT 2wk (MPT measured at week 2).

SECONDARY OUTCOMES:
Severity of pain | week 0 to week 12
  Pain was measured by a numerical rating scale (NRS), with 0 symbolizing no pain and 10 symbolizing the worst pain one could imagine.
Sleep | week 0 to week 12
  The quality of sleep was measured by Athens Insomnia Scale.
Depression and anxiety | week 0 to week 12
  Depression was measured by Patient Health Questionnaire-9. Anxiety was measured by a Generalized Anxiety Disorder-7 item scale.
Life quality | week 0 to week 12
  The quality of life was measured by Short Form 36 Health Survey.

IPD SHARING:
Plan to Share IPD: No